CLINICAL TRIAL: NCT05496166
Title: Comparing the Efficiency Between Surgery and Radiotherapy After SHR-1316 (Adebrelimab) and Platinum-containing Doublet Induction Therapy for Limited-stage Small Cell Lung Cancer: a Randomized, Controlled, Open-label, Single-center Phase III Clinical Trial
Brief Title: The Efficiency of Surgery and Radiotherapy After SHR-1316 (Adebrelimab) and Platinum-containing Doublet Induction Therapy for Limited-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Peng Zhang, associate professor of medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-015
Record Dates: First submitted 2022-07-27; First posted 2022-08-11 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-08

CONDITIONS: Limited Stage Small Cell Lung Cancer
Keywords: LD-SCLC; surgery; radiotherapy; neoadjuvant chemoimmunotherapy
MeSH Terms: interventions — Drug Therapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery group (Experimental): SHR-1316+chemotherapy+surgery
  Interventions: Combination Product: chemotherapy and SHR-1316(Adebrelimab) comnined with surgery or radiotherapy
- radiotherapy group (Active Comparator): SHR-1316+chemotherapy+radiotherapy
  Interventions: Combination Product: chemotherapy and SHR-1316(Adebrelimab) comnined with surgery or radiotherapy

INTERVENTIONS:
Combination Product: chemotherapy and SHR-1316(Adebrelimab) comnined with surgery or radiotherapy — Induction treatment stage: SHR-1316(Adebrelimab)，20mg/kg,+Cisplatin 75mg/m2, d1+ etoposide 100mg/m2, d1,d2,d3, q3w, iv, 4 cycles. Patients who are able to receive surgery after assessed by two surgons would receive surgery or radiotherapy randomly. Adjuvant/ maintenance treatment stage: SHR-1316，20mg/kg, iv, q3w,up to 1 year

SUMMARY:
To compare the efficiency between surgery and radiotherapy after SHR-1316 (Adebrelimab)and platinum-containing doublet induction therapy for limited-stage small cell lung cancer

DETAILED DESCRIPTION:
1.1 Main purpose To compare the efficiency between surgery and radiotherapy after therapy with SHR-1316 and chemotherapy for limited-stage small cell lung cancer according to progression-free survival (PFS) 1.2 Secondary Purpose The incidence of adverse events (AEs) during treatment was assessed to identify the safety of SHR-1316 and chemotherapy combined with surgery or radiotherapy according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

To evaluate the pathological response rate (MPR and PCR) of the surgical population after neoadjuvant therapy with SHR-1316 and chemotherapy for operable LD-SCLC according to the evaluation criteria of pathological response after neoadjuvant therapy recommended by the International Association for the Study of Lung Cancer (IASLC); To evaluate the overall survival (OS) of patients with limited-stage small cell lung cancer after therapy with SHR-1316 and chemotherapy combined with surgery or radiotherapy To evaluate the recurrence-free survival (RFS) in patients with limited-stage small cell lung cancer who received neoadjuvant SHR-1316 and chemotherapy combined with surgery; To evaluate the duration of response (DOR) in patients with limited-stage small cell lung cancer after SHR-1316 and chemotherapy combined with surgery or radiotherapy according to RECIST v1.1 To identify the impact on the health-related quality of life (HRQoL), mood, symptoms, sleep, etc. of patients undergoing surgery and radiotherapy after therapy with SHR-1316 and chemotherapy according to the Pulmonary Hospital Psychological Assessment Scale; 1.3 Exploratory Purpose To explore potential predictive biomarkers in archived and/or fresh tumor tissue and/or blood (or blood derivatives), including but not limited to programmed cell death protein ligand 1 (PD-L1) expression as determined by immunohistochemistry (IHC), gene expression profile (GEP), tumor mutational burden (TMB), tumor-infiltrating immune cell changes, etc., to evaluate the association of these markers with the study of treatment response or resistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* after signing informed consent;
* Aged 18-70;
* Histologically or cytologically confirmed SCLC, imaging examination and other confirmed limited-stage small cell lung cancer, and without previous treatment;
* For clinical stage IIB-III, all patients should have clear lymph node pathology by EBUS to exclud occult lymph node metastasis.
* Two thoracic surgeons assessed thar it would be able to achieve radical surgery or R0 resection after 4 cycles of treatment. Surgical approaches include lobectomy, sleeve resection and pneumonectomy
* ECOG performance status score 0-1 points;
* With a life expectancy of at least 12 weeks;
* At least one measurable tumor
* With normal Other major organs (liver, kidney, blood system, etc.) function:

Absolute neutrophil count (ANC) ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥90 g/L. Note: Patients should not receive blood transfusion or growth factor support within ≤ 14 days before blood collection during the screening period;

- International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × upper limit of normal (ULN); Activated partial thromboplastin time (APTT) ≤ 1.5×ULN; Serum total bilirubin ≤ 1.5×ULN (total bilirubin in patients with Gilbert syndrome must be <3×ULN); Aspartate and alanine aminotransferase (AST and ALT) ≤2.5×ULN, or AST and ALT ≤5×ULN in patients with liver metastases

* Female patients of childbearing potential must voluntarily use highly effective contraception during the study period until ≥ 120 days after the last dose of chemotherapy or SHR-1316, whichever is later, and have ≤ 7 days of urine or Serum pregnancy test results are negative;
* Unsterilized male patients must voluntarily use highly effective contraception during the study period until ≥120 days after the last dose of chemotherapy or SHR-1316, whichever is later.

Exclusion Criteria:

* Received any systemic anticancer therapy, including surgery, local radiotherapy, cytotoxic drug therapy, targeted drug therapy, and experimental therapy;
* Patients with other malignancies within five years prior to the start of the trial;
* Combined with unstable systemic diseases, such as uncontrolled hypertension, severe arrhythmia, etc;
* With active, known or suspected autoimmune disease, or autoimmune paraneoplastic syndrome requiring systemic therapy;
* Allergy to the test drug;
* Have or currently have interstitial lung disease;
* Coexisting with HIV infection or active hepatitis;
* Patients who have undergone other major surgery or severe trauma within 2 months before the start of the trial;
* Pregnant or breastfeeding women;
* Those who suffer from neurological diseases or mental illnesses who cannot cooperate;
* Other reasons that investigators deem inappropriate for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years
  It refers to the time from the first administration of SHR1316 in this study to the disease progression or death (including any cause of death in the case of no progression) , regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.

SECONDARY OUTCOMES:
incidence of adverse events | through study completion, an average of 1.5 years
  The frequency of severe adverse events as assessed by CTCAE 5.0 from the participants enrolling to 90 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
pathological response | up to 5 months
  To evaluate the pathological response rate (major pathological response and complete pathological response) of the surgical population after neoadjuvant therapy with SHR-1316 and chemotherapy for operable LD-SCLC according to the evaluation criteria of pathological response after neoadjuvant therapy recommended by the International Association for the Study of Lung Cancer (IASLC)
objective response rate | through study completion, an average of 1.5 years
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation
overall survival | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
recurrence free survival | up to 60 months
  It is defined as the time from enrollment to recurrence in patients who received surgery
the duration of response(DOR) | up to 60 months
  the time from the date when the response criteria of complete response or partial response is first met to the date of progression/relapse or death.

OTHER OUTCOMES:
biological predicted markers | through study completion, an average of 1.5 years
  to explore potential predictive biomarkers in archived and/or fresh tumor tissue and/or blood (or blood derivatives), including but not limited to programmed cell death protein ligand 1 (PD-L1) expression as determined by immunohistochemistry (IHC), gene expression profile (GEP), tumor mutational burden (TMB), tumor-infiltrating immune cell changes, etc., to evaluate the association of these markers with the study of treatment response or resistance mechanisms

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shang'ai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No